CLINICAL TRIAL: NCT02661087
Title: MONOBISY: Randomized Controlled Trial Comparing Intra Uterine Synechiae Occurence Using Bipolar Energy Compared With Monopolar Energy in Myoma Resection on Women Having Menorraghia and/or Infertility
Brief Title: Comparing Intra Uterine Synechiae Occurence Using Bipolar Energy Compared With Monopolar Energy in Myoma Resection on Women Having Menorraghia and/or Infertility
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator departure
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Andre Nazac, Head of Clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUB-Monobisy
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Symptomatic Submucosal Myoma
Keywords: submucosal myoma; hysteroscopic resection; bipolar energy; monopolar energy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar energy (Experimental): Hysteroscopic resection of symptomatic sub mucosal myomas with the use of bipolar energy
  Interventions: Procedure: Hysteroscopic resection with bipolar energy
- Monopolar energy (Active Comparator): Hysteroscopic resection of symptomatic sub mucosal myomas with the use of monopolar energy
  Interventions: Procedure: Hysteroscopic resection with monopolar energy

INTERVENTIONS:
Procedure: Hysteroscopic resection with bipolar energy — Hysteroscopic resection with bipolar energy
  Arms: Bipolar energy
Procedure: Hysteroscopic resection with monopolar energy — Hysteroscopic resection with monopolar energy
  Arms: Monopolar energy

SUMMARY:
Since the development in the last few years of the bipolar energy in the surgery by hysteroscopy, the hysteroscopic treatment of the submucosal uterine myoma can be performed by use of either monopolar or bipolar current.

It seems that the use of the bipolar energy decreases the rate of adhesions but prospective data on the adhesion rate and fertility after the use of bipolar energy during the surgery are poor, and there is currently no recommendation as to the choice of technique to use. The main purpose of this study is to compare the rate of uterine adhesions six weeks after the surgical hysteroscopic treatment of uterine submucosal myoma, by using monopolar or bipolar energy. The pregnancy and spontaneous miscarriage rate will also be evaluated.

DETAILED DESCRIPTION:
Uterine fibroids are detected in many cases of excessive bleeding or consultation for primary or secondary infertility. When they are of the submucosal type, they require a surgical treatment by hysteroscopy. The hysteroscopic resection of submucosal fibroids described by Neuwirth and Amin in 1976 allowed to reduce the morbidity, the length of hospital stay and the cost of the therapeutic treatment, with a satisfactory rate of functional successes.

The surgical hysteroscopic treatment of symptomatic submucosal myoma was performed initially by a monopolar endoscopic resection. This required a resection using glycine as a distension medium, essential for the conduction of monopolar current.

Complications proper to the monopolar resection have been described and are now well known. The first specific complication is the TURP syndrome, linked to the reabsorption of the glycine byproducts of the distensium medium. It can cause hyponatremia and lead to a cerebral edema. This complication can be prevented by limiting the duration of the intervention to 45 minutes and constantly monitoring the input-output balance.

The second specific complication is related to the diffusion of heat that can damage to surrounding healthy tissue and increase the risk of uterine adhesions. These adhesions are the source of menstrual disorders like hypomenorrhea or amenorrhea, infertility or a recurrent miscarriages.

For over 20 years, several approaches have been proposed to reduce the occurrence of postoperative adhesions. However, their results are either not convincing, either in need of confirmation.

Since several years, the use of the bipolar energy for hysteroscopic resection has been developped.The advantage of this technique is to avoid glycine as distension medium and use saline instead, hereby significantly reducing the risk of hyponatremia. It especially gives a smaller heat diffusion, hereby limiting the damage to the healthy tissues nearby.

Although hysteroscopic bipolar resection of submucosal fibroids is now a routine technique, there are to this date no studies in the literature comparing the use of monopolar and bipolar energy in the hysteroscopic myomectomy.

The main objective of this study is to compare the rate of adhesions after resection of uterine myomas, with the use of bipolar versus monopolar current. The secondary objective is to evaluate the impact on subsequent fertility through the number of pregnancies and miscarriages.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic (menorrhagia or primary/secondary infertility) with pregnancy wishes
* One submucosal myoma, type 0 to Type II, accessible to a hysteroscopic surgery

Exclusion Criteria:

* Several submucosal myomas
* Pregnant woman
* Patient under anticoagulating treatment (anti-vitamin K-type)
* Patient with a malignant endometrial pathology
* Patient having one or more endo-uterine synechiae
* Myoma larger than 5 cm
* Uterine malformation
* Active infection, not healed
* Refusal to participate in the Protocol

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
uterine adhesions rate | 6 weeks after surgery
  The main goal of this study is to compare the rate of uterine adhesions six weeks after the hysteroscopic surgical treatment of sub mucosal uterine myomas, in a group where bipolar energy is used versus a group where monopolar energy is used during the surgery. Outcome measured at the diagnostic hysteroscopic visit, 6 weeks after surgery.

SECONDARY OUTCOMES:
Pregnancy rate | 18 months after surgery
  Number of evolutive pregnancies - phone contact 18 months after surgery
Spontaneous abortion rate | 18 months after surgery
  Number of spontaneous abortions - phone contact 18 months after surgery
Surgery duration | From the entry to the exit of the hysteroscope from the body. Ambulatory surgery, max 1 day
  Duration of the surgical intervention
Per-surgery complications rate | From the entry to the exit of the hysteroscope from the body. Ambulatory surgery, max 1 day
  Complications rate during the surgery duration
Post-surgery complications rate | 6 weeks after surgery
  Post-surgery complications rate, measured at the diagnostic hysteroscopic visit performed 6 weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: André Nazac, MD, Principal Investigator — CHU Brugmann
Locations (2):
- CHU Brugmann, Brussels, Belgium
- CHU Bicêtre, Kremlin Bicêtre, Le Kremlin-Bicêtre, France

REFERENCES:
- [Background] Neuwirth RS, Amin HK. Excision of submucus fibroids with hysteroscopic control. Am J Obstet Gynecol. 1976 Sep 1;126(1):95-9. doi: 10.1016/0002-9378(76)90471-3. PMID 961753
- [Background] Valle RF, Sciarra JJ. Intrauterine adhesions: hysteroscopic diagnosis, classification, treatment, and reproductive outcome. Am J Obstet Gynecol. 1988 Jun;158(6 Pt 1):1459-70. doi: 10.1016/0002-9378(88)90382-1. PMID 3381869
- [Background] Jewelewicz R, Khalaf S, Neuwirth RS, Vande Wiele RL. Obstetric complications after treatment of intrauterine synechiae (Asherman's syndrome). Obstet Gynecol. 1976 Jun;47(6):701-5. PMID 934560
- [Background] Taskin O, Sadik S, Onoglu A, Gokdeniz R, Erturan E, Burak F, Wheeler JM. Role of endometrial suppression on the frequency of intrauterine adhesions after resectoscopic surgery. J Am Assoc Gynecol Laparosc. 2000 Aug;7(3):351-4. doi: 10.1016/s1074-3804(05)60478-1. PMID 10924629
- [Background] Acunzo G, Guida M, Pellicano M, Tommaselli GA, Di Spiezio Sardo A, Bifulco G, Cirillo D, Taylor A, Nappi C. Effectiveness of auto-cross-linked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic adhesiolysis: a prospective, randomized, controlled study. Hum Reprod. 2003 Sep;18(9):1918-21. doi: 10.1093/humrep/deg368. PMID 12923149
- [Background] Guida M, Acunzo G, Di Spiezio Sardo A, Bifulco G, Piccoli R, Pellicano M, Cerrota G, Cirillo D, Nappi C. Effectiveness of auto-crosslinked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic surgery: a prospective, randomized, controlled study. Hum Reprod. 2004 Jun;19(6):1461-4. doi: 10.1093/humrep/deh238. Epub 2004 Apr 22. PMID 15105384
- [Background] Vilos GA, Abu-Rafea B. New developments in ambulatory hysteroscopic surgery. Best Pract Res Clin Obstet Gynaecol. 2005 Aug;19(5):727-42. doi: 10.1016/j.bpobgyn.2005.06.012. Epub 2005 Aug 26. PMID 16126460
- [Background] Touboul C, Fernandez H, Deffieux X, Berry R, Frydman R, Gervaise A. Uterine synechiae after bipolar hysteroscopic resection of submucosal myomas in patients with infertility. Fertil Steril. 2009 Nov;92(5):1690-3. doi: 10.1016/j.fertnstert.2008.08.108. Epub 2008 Oct 19. PMID 18937941